CLINICAL TRIAL: NCT02967328
Title: A Multi-Center Prospective Blind Study of RP% Measurement by Flow Cytometry in the Diagnosis of Primary Immune Thrombocytopenia
Brief Title: RP% Measurement by FCM as a Diagnostic Test for ITP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Jinan Central Hospital (Other); Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Other Study IDs: ITP-Reticulated Platelets
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Immune Thrombocytopenia
Keywords: Reticulated Platelets; Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Inosine Triphosphate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- RP% Measurement by FCM as a Diagnostic Test for ITP: The investigators are undertaking a multi-center, prospective blind trial of 500 adults with thrombocytopenic disorders with a platelet count less than 60000/uL from 4 medical centers in China. In brief, 15 ul aliquots of anti-coagulated whole blood were incubated for 70 min with 5 ul of phycoerythrin-conjugated anti-CD42b monoclonal antibody (BD Pharmingen, Tokyo, Japan) and 1 ml of thiazole orange (Retic-COUNT; Becton-Dickinson, San Jose, CA, USA) diluted 10 times by phosphate-buffered saline. RP% was analyzed on a flow cytometer (FACScan, Becton-Dickinson) by measuring 10,000 events in the CD42b-positive fraction.
  Interventions: Other: RP% Measurement by FCM as a Diagnostic Test for ITP

INTERVENTIONS:
Other: RP% Measurement by FCM as a Diagnostic Test for ITP

SUMMARY:
Immature platelets-also termed reticulated platelets (RP)-are platelets newly released into the circulation, and have been associated with a variety of pathological bleeding events including primary immune thrombocytopenia (ITP). They can be assessed by flow cytometry (FCM) after staining with thiazole orange (TO) at low concentration and expressed as a fraction of the total platelet count (RP%). The diagnosis of primary ITP is based on differential diagnosis and the measurement of RP% can serve as an alternative diagnostic test that are useful in daily practice. Our study aimed at distinguishing primary ITP from other thrombocytopenic disorders, especially aplstic (hypoplastic) or chemotherapy-induced thrombocytopenia by FCM. The sensitivity and specificity of the assay as well as agreement between RP% measurement and monoclonal antibody-specific immobilization of platelet antigen (MAIPA) were analyzed accordingly.

DETAILED DESCRIPTION:
The investigators are undertaking a multi-center, prospective blind trial of 500 adults with thrombocytopenic disorders with a platelet count less than 60*10^9/L from 4 medical centers in China. In brief, 15 μl aliquots of anti-coagulated whole blood were incubated for 70 min with 5 μl of phycoerythrin-conjugated anti-CD42b monoclonal antibody (BD Pharmingen, Tokyo, Japan) and 1 ml of thiazole orange (Retic-COUNT; Becton-Dickinson, San Jose, CA, USA) diluted 10 times by phosphate-buffered saline. RP% was analyzed on a flow cytometer (FACScan, Becton-Dickinson) by measuring 10,000 events in the CD42b-positive fraction.

Clinical information of all participants including gender, age, platelet count and definitive diagnosis were recorded by an exclusive investigator. RP% results were revealed at the end of recruitment and after all FCM measurements were completed. The agreement between clinical diagnosis and RP% results were analyzed to identify primary ITP.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated adult patients of both gender between the ages of 18 and 75 years
2. Each participant showed a platelet count 60*10^9/L, with or without bleeding manifestations
3. Thrombocytopenic disorders including autoimmune-mediated, aplastic (hypoplastic) or chemotherapy-induced thrombocytopenia

Exclusion Criteria:

1. Received high-dose steroids or IVIG within 3 weeks prior to the test
2. Received second-line ITP-specific treatments (eg, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) within 3 months prior to the test
3. Current HIV infection, hepatitis B virus or hepatitis C virus infections
4. Severe medical condition (liver and kidney function impairment). Unstable cardiovascular disease or uncontrolled hypertension.
5. Patients who are deemed unsuitable for the study by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 adults with thrombocytopenic disorders with a platelet count less than 60000/uL from 4 medical centers in China.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Total platelet count (RP%) | The day upon enrollment
  We defined an upper limit for healthy control subjects as mean + 3SD in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Result] Sakuragi M, Hayashi S, Maruyama M, Kabutomori O, Kiyokawa T, Nagamine K, Kato H, Kashiwagi H, Kanakura Y, Tomiyama Y. Clinical significance of IPF% or RP% measurement in distinguishing primary immune thrombocytopenia from aplastic thrombocytopenic disorders. Int J Hematol. 2015 Apr;101(4):369-75. doi: 10.1007/s12185-015-1741-0. Epub 2015 Jan 25. PMID 25618218
- [Result] Ibrahim H, Nadipalli S, Usmani S, DeLao T, Green L, Kleiman NS. Detection and quantification of circulating immature platelets: agreement between flow cytometric and automated detection. J Thromb Thrombolysis. 2016 Jul;42(1):77-83. doi: 10.1007/s11239-016-1338-3. PMID 26831482